CLINICAL TRIAL: NCT03423888
Title: Acceptability of High-flow Nasal Oxygen to Relieve Dyspnea in Palliative Care: Pilot Study
Brief Title: High-flow Nasal Oxygen in Palliative Care: Pilot Study
Acronym: OXYPALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/17/0351; 2017-A03377-46 (Other: Id-RCB number)
Record Dates: First submitted 2018-01-26; First posted 2018-02-06 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Dyspnea
Keywords: Dyspnea; palliative care; high-flow nasal oxygen; pilot study
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-flow nasal oxygen (Experimental)
  Interventions: Device: high-flow nasal cannula oxygen therapy (HNFC)

INTERVENTIONS:
Device: high-flow nasal cannula oxygen therapy (HNFC) — Set up of high-flow nasal oxygen for patient with dyspnea for a respiratory disease without possibility of curative care. Patients who require a treatment by oxygen are included.
  After 7 days of treatment, acceptability is evaluated by the duration of use of HNFC.

SUMMARY:
In palliative care, the relief of the dyspnea is necessary. Medications for the reduction of dyspnea have side effects. High-flow nasal cannula oxygen therapy (HFNC) is a new way to deliver oxygen. Investigators hypothesize that HNFC is an acceptable technic for the patient with dyspnea in palliative care.

A pilot study with 30 patients will be conducted. Acceptability of HNFC will be studied by the time of use by patients of the HNFC during one week. The effectiveness of HNFC in relieving dyspnea will be studied using Borg scale.

DETAILED DESCRIPTION:
Pilot study for acceptability of high flow nasal cannula oxygen therapy in palliative care Population: 30 patients in palliative care (for lung cancer, terminal respiratory failure) who suffer from dyspnea and have oxygen therapy. Patients with curative care are excluded and patients who require non invasive ventilation.

An oral consent is asked.

Primary objective: acceptability of HNFC in patients with dyspnea in palliative care during one week

Secondary objectives:

* Tolerance of HNFC at short term (1h and 24h) and long term (7 days) after initiation of HNFC
* Efficiency of HNFC at short term

Primary outcome: duration of use of the HNFC during 7 days

Secondary outcome:

* Tolerance: noise of the system of HNFC, side effects of high flow (nasal dryness..)
* Efficiency: evaluation of dyspnea by Borg scale and measure of respiratory rate and saturation of oxygen one hour after initiation of HNFC

ELIGIBILITY:
Inclusion Criteria:

* Patient followed for respiratory failure with palliative care and :
* More than 18 years old
* Dyspnea related to a respiratory disease
* Hypoxemia requiring the introduction of more than 4 liters of oxygen for a sp02 > 90%
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient less than 18 years old
* Patient with guardianship, trusteeship
* No consent for participation at the study
* Project of curative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Acceptability of HNFC in patients with dyspnea in palliative care during one week | 7 days
  Duration of use of HNFC: nurses will set up the device to the patient who can withdraw it at any time. It will then be noted the stop time and recovery of the device for a week, which will know the time of use and acceptability. If the patient wishes to permanently stop the use of the device, the stop time will be raised.

SECONDARY OUTCOMES:
Efficiency of high-flow nasal oxygen in palliative care with dyspnea | At short term: one hour after the initiation and at long term: 24h and seven days after the start
  Evaluation of dyspnea with the Borg scale. The Borg scale is a scale containing 10 proposals ranging in increasing order of severity (from no gene at all to extremely embarrassed) that will allow the patient to grading his respiratory gene.
Efficiency of high-flow nasal oxygen in palliative care with Sp02 | At short term: one hour after the initiation and at long term: 24h and seven days after the start
  Evaluation of Sp02 using transcutaneous oximeter
Efficiency of high-flow nasal oxygen in palliative care with respiratory rate | At short term: one hour after the initiation and at long term: 24h and seven days after the start
  Evaluation of respiratory rate

OTHER OUTCOMES:
Tolerance of high-flow nasal oxygen in palliative care | At short term: one hour after the initiation and at long term: 24h and seven days after the start
  Side effects (nasal dryness, nasal lesion) and noise with an numerical scale graduated from 0 to 10 (0 for no noise to 10 very noisy)

CONTACTS AND LOCATIONS:
Overall Officials: Marion DUPUIS, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hospital LARREY, CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No